CLINICAL TRIAL: NCT01645748
Title: Multicenter Phase II Study of Weekly Docetaxel, Cisplatin, and S-1 (TPS) Induction Chemotherapy in Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Docetaxel, Cisplatin, and S-1 (TPS) Induction Chemotherapy in Locally Advanced Head and Neck Cancer
Acronym: TPSHNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chungbuk National University (Other); Chonbuk National University (Other); Chungnam National University (Other)
Responsible Party: Principal Investigator, Sang-Hee Cho, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUHH-MO-02; CNUHH (Other Grant/Funding Number: Jeil Pham)
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; docetaxel; cisplatin; S-1
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — S 1 (combination); titanium silicide; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1, induction chemotherapy (Experimental): Cisplatin and 5-FU is the standard treatment for patients with head and neck cancer. Recently,docetaxel was used into CF, and it showed the prolongation of survival. Oral 5-FU showed similar or enhanced response rate, safety than intravenous 5-FU. S-1 showed promising preliminary result in combination with cisplatin in head and neck cancer. In patients with gastric cancer, phase I study of S-1, docetaxel and cisplatin combination chemotherapy was reported and the recommended doses were 40mg/m2 bid, 60mg/m2 (D1) and 60mg/m2 (D1), respectively. And weekly docetaxel can reduce adverse events compared to 3 week regimen. The aim of this study was to evaluate the efficacy and safety of weekly docetaxel, cisplatin and S-1 combination chemotherapy
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — S-1 is an oral fluoropyrimidine derivative, based on the concept of biochemical modulation. It consists in a molar ratio of 1:0.4:1: tegafur, a prodrug that is slowly metabolized to 5-fluorouracil; gimeracil, which reversibly inhibits dihydropyrimidine dehydrogenase. In patients with advanced gastric cancer, phase I study of S-1, docetaxel and cisplatin combination chemotherapy was reported and the recommended doses were 40mg/m2 bid (D1-D14), 60mg/m2 (D1) and 60mg/m2 (D1), respectively.
  Other Names: TS-1
Drug: S-1 — Chemotherapy was comprised of docetaxel 30 mg/m2 on days 1 and 8, cisplatin 60 mg/m2 on day 1, and S-1 70 mg/m2 on days 1 to 14, with the regimen repeated every 21 days
  Other Names: TS-1
Drug: S-1 — In patients with advanced gastric cancer, phase I study of S-1, docetaxel and cisplatin combination chemotherapy was reported and the recommended doses were 40mg/m2 bid (D1-D14), 60mg/m2 (D1) and 60mg/m2 (D1), respectively. Another phase II study of TPS as induction chemotherapy for locally advanced HNSCC was determined to be 70/70/60 mg∙m2/d every 3 weeks. However, the rate of grade 3-4 neutropenia was 75% at this recommended dose. To reduce the hematologic toxicities, we used the docetaxel weekly. Therefore following regimen was evaluated in this study; docetaxel 30 mg/m2 (D1, D8), cisplatin 60mg/m2 (D1), S-1 70mg/m2 (D1-D14) every 3 weeks.
  Other Names: TS-1; docetaxel; cisplatin

SUMMARY:
The purpose of this study was to evaluate the tolerability and efficacy of a combination of weekly docetaxel, cisplatin, and S-1 (weekly TPS) as induction chemotherapy in patients with locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
Combination chemotherapy with cisplatin and fluorouracil (CF) is the standard treatment for patients with locally advanced squamous cancer of the head and neck. CF chemotherapy has been reported to increase survival and disease free survival in patients with unresectable disease when given before definitive radiotherapy, showing overall response rate as 75-85% including of CR rate of 25-35%. To improvement of treatment, docetaxel was incorporated into CF as induction treatment and it showed the prolongation of progression free survival and overall survival in large scale of randomized phase III trials, therefore triple combination induction regimen would be standard treatment in advanced head and neck cancer. Recently, the introduction of oral fluoropyrimidine showed similar or enhanced response rate, also favorable safety and convenience than intravenous fluoropyrimidine in advanced gastric cancer. Of the oral fluoropyrimidines, S-1 showed promising preliminary result in combination chemotherapy with cisplatin in head and neck cancer. In patients with advanced gastric cancer, phase I study of S-1, docetaxel and cisplatin combination chemotherapy was reported and the recommended doses were 40mg/m2 bid, 60mg/m2 (D1) and 60mg/m2 (D1), respectively. Therefore, the aim of this study was to evaluate the efficacy and safety of docetaxel, cisplatin and S-1 combination chemotherapy according to above dosage.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced stage III or IV squamous cell carcinoma of the larynx, oropharynx, or hypopharynx
* ≥18 years old
* absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL
* serum bilirubin <2.0 mg/dL
* creatinine <1.5 mg/dL
* serum transaminase levels less than twice the upper limit of normal

Exclusion Criteria:

* received previous chemotherapy
* another malignancy
* current or history of distant metastasis
* history of clinically significant cardiac disease within 6 months
* active serious infection
* nasopharyngeal carcinoma
* psychiatric illness that would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Response rate was evaluated 1 months after completion of CCRT
  After completion of CCRT, response rate was assessed. Patients underwent examination by an otolaryngologist, CT or MRI imaging of the primary tumor and neck. A biopsy of the primary site was recommended if possible. Tumor response was assessed according to the RECIST. For all patients with complete response (CR) on physical examination and CT or MRI scan, PET scan was performed for confirmation at 1 month after CT or MRI confirmation.

SECONDARY OUTCOMES:
Safety | From initiation of induction chemotherapy up to 18 weeks
  Number of participants with adverse events as a measure of safety according to NCI-CTC version 3.0 was checked every 3 weeks up to 18 weeks.
Progression free survival | From initiation of treatment up to 2 years
  Progression free survival means that the time from date of initiation of treatment until the date of first documented progression. Patients who completed treatment were followed by physician examination and CT or MRI scanning every 3 months for 1 year and then these checkup was done every 6 months for another one year.
Overall survival | From initiatin of treatment up to 2 years
  Overall survival means that the time from initiation of treatment until the date of death from any cause up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hee Cho, M.D.Ph.D., Principal Investigator — CNUHH
Locations (1):
- Chonnam National University Hwasun Hospital, Gwangju, Jeollanamdo, South Korea

REFERENCES:
- [Derived] Bae WK, Hwang JE, Shim HJ, Cho SH, Lee KH, Han HS, Song EK, Yun HJ, Cho IS, Lee JK, Lim SC, Chung WK, Chung IJ. Multicenter phase II study of weekly docetaxel, cisplatin, and S-1 (TPS) induction chemotherapy for locally advanced squamous cell cancer of the head and neck. BMC Cancer. 2013 Mar 6;13:102. doi: 10.1186/1471-2407-13-102. PMID 23497365